CLINICAL TRIAL: NCT02368119
Title: A PHASE IB, DOUBLE-BLIND, CLINICAL TRIAL TO EVALUATE THE SAFETY, TOLERABILITY AND IMMUNOGENICITY OF TWO DIFFERENT DOSAGE LEVELS OF EBOLA CHIMPANZEE ADENOVIRUS VECTOR VACCINE "VRC-EBOADC069-00-VP (cAd3-EBO)" AND THE HETEROLOGOUS PRIME-BOOST CANDIDATE VACCINE REGIMEN OF cAD3-EBO FOLLOWED BY MVA-VECTORED VACCINE IN HEALTHY ADULTS, 18-65 YEARS OF AGE, IN BAMAKO, MALI
Brief Title: Ebola CVD-Mali #2000 (Bivalent) VRC-EBOAdc069-00-vp (cAd3-EBO)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Milagritos Tapia, Assistant Professor, Pediatrics & Infectious Tropical Diseases, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HP-00062548
Record Dates: First submitted 2015-02-05; First posted 2015-02-20 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Ebola Virus Disease; Hemorrhagic Fever
MeSH Terms: conditions — Hemorrhagic Fever, Ebola; Hemorrhagic Fevers, Viral

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): VRC-EBOADC069-00 VP (cAd3-EBO bivalent (Zaire plus Sudan) vaccine (2 x 10(10) vp (n=10) or VRC-EBOADC069-00 VP (cAd3-EBO bivalent (Zaire plus Sudan) vaccine (2 x 10(11) vp (n=10). Randomization to booster of MVA-EbolaZ or PBS placebo will be completed 4 to 16 weeks after priming dose.
  Interventions: Biological: VRC-EBOADC069-00-vp; Biological: MVA-EbolaZ; Other: Placebo
- Group 2 (Experimental): VRC-EBOADC069-00 VP (cAd3-EBO bivalent (Zaire plus Sudan) vaccine (2 x 10(10) vp (n=20) or VRC-EBOADC069-00 VP (cAd3-EBO bivalent (Zaire plus Sudan) vaccine (2 x 10(11) vp (n=20). Randomization to booster of MVA-EbolaZ or PBS placebo will be completed 4 to 16 weeks after priming dose.
  Interventions: Biological: VRC-EBOADC069-00-vp; Biological: MVA-EbolaZ; Other: Placebo

INTERVENTIONS:
Biological: VRC-EBOADC069-00-vp — IM Injection of cAd3-EBO bivalent (Zaire plus Sudan) vaccine (2 x 10(10) vp)
  Other Names: cAd3-EBO at 2x10(10) vp
Biological: VRC-EBOADC069-00-vp — IM Injection of cAd3-EBO bivalent (Zaire plus Sudan) vaccine (2 x 10(11) vp)
  Other Names: cAd3-EBO at 2x10(11) vp
Biological: MVA-EbolaZ — IM injection of MVA-EbolaZ vaccine
Other: Placebo — IM injection injection of Phosphate Buffered Saline

SUMMARY:
Ebola virus causes an infection known as Ebola virus disease (EVD). This it is generally a severe disease which can also lead to death. The 2014 outbreak of EVD in West Africa is the largest ever. Researchers want to develop a vaccine to prevent Ebola infection.

This study will assess the safety of a single dose of the bivalent Ebola Zaire candidate vaccine VRC-EBOADC069-00-VP (cAD3-EBO) when administered to healthy Malian adult volunteers, age 18-65 years (mostly health care workers and other front line workers [e.g., individuals who incinerate contaminated materials]), at one of 2 dosage levels, 2.0 x 10(10) vp or 2 x 10(11) vp. It is impossible for someone to get an Ebola infection from this vaccine.

Heterologous booster dose allocation - Each participant will be offered the opportunity to be included in the booster step of this study. After obtaining consent and the additional review of pertinent medical history, participants in each group will be randomized to receive the candidate booster vaccine, MVA-EbolaZ or placebo.

This will be the first clinical trial in Mali with bivalent cAd3-based Ebola vaccine and the first where the dosage level contains > 10(11) vp. It follows completion of a Phase Ib trial in Malian health care workers that tested three dosage levels of monovalent cAd3-EBO Z vaccine. The data generated in West Africans (Mali) on the tolerability and immunogenicity of the bivalent vaccine will be compared to clinical and immunologic responses documented in in parallel studies in East African subjects (Uganda) and North American subjects (NIH, Bethesda, MD, USA).

Objectives:

* To see if an Ebola vaccine is safe and to study immune responses to it.
* To study the effect of the MVA-EbolaZ booster on the immune response

Eligibility:

- Healthy adults ages 18-65.

DETAILED DESCRIPTION:
This is a phase 1B, double-blind, randomized study to examine the safety, tolerability and immunogenicity of two different dosage levels of investigational Ebola vaccine.

The vaccine is a recombinant chimpanzee adenovirus Type 3-vectored Ebolavirus vaccine (cAd3-EBO), VRC-EBOADC069-00-VP. The vaccine encodes wild type (WT) glycoproteins (GP) from Zaire and Sudan species of Ebola virus. The primary objective is to assess the safety of a single dose intramuscular injection of the bivalent vaccine at one of 2 dosage levels, 2.0 X 10(10) vp or 2 x 10(11) vp and to assess the safety of the heterologous prime boost regimen of cAd3-EBO followed by MVA-EbolaZ or Phosphate Buffered Saline (PBS) placebo. A secondary objective is to assess the immunogenicity generated by 2 different dosage levels of the bivalent Ebola candidate vaccine.

Enrolment of Group 1 participants:

The first 20 Malian volunteers will be vaccinated in a staggered fashion. For safety reasons, the first 10 Malian subjects to receive a vaccine dose in Group 1 will be vaccinated on day 1 and we will wait 24 hours before vaccinating 10 subsequent volunteers. After these 20 volunteers in Group 1 have been vaccinated and followed up for 7 days, an interim safety review (ISR1) will be performed by the DSMB. Enrolment of subjects into Group 2 will commence only after the DSMB has assessed the data and indicated that it is safe to do so.

Half of Group 1 participants will be randomly assigned to receive the low dose and the remaining 10 will be randomized to receive the high dose.

Enrolment of Group 2 participants:

The 40 subjects in Group 2 will be accrued as rapidly as possible. The 40 Malian volunteers in Group 2 will be vaccinated over several days to limit wastage of the available doses of cAd3 EBO. As a result, a proposed scheme would be 10 per vaccination day. This could be adjusted as needed to limit wastage but no more than 20 participants would be vaccinated in 1 day. After the total of 40 volunteers in Group 2 have been vaccinated and followed up for 7 days, an interim safety review (ISR2) will be performed by the DSMB.

Prime Boost Vaccine Randomization 4-16 weeks after priming dose: Each participant will be offered the opportunity to be included in the booster step of this study. After obtaining consent and the additional review of pertinent medical history, participants in each group will be randomized to receive the candidate booster vaccine, MVA-EbolaZ or PBS placebo

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 65 years
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* For females only, willingness to practice continuous effective contraception (see section 6.4.3) during the study and a negative urine pregnancy test on the day(s) of screening and vaccination
* Agreement to refrain from blood donation during the course of the study
* Provide written informed consent

Laboratory criteria within 30 days prior to enrollment:

* Hemoglobin ≥ 11.0 g/dL for women; ≥12.5 g/dL for men.
* White blood cells (WBC) = 2,500-11,000 cells/mm3.
* Neutrophil count = 1200 - 7000 cells/mm3
* Lymphocyte count ≥ 800 cells/mm3
* Eosinophil count = 0 - 500 cells/mm3
* Platelets = 125,000 - 400,000/mm3
* Alanine aminotransferase (ALT) = 10-45 IU/L
* Serum creatinine = 54-145 umol/L.
* HIV-uninfected as evidenced by a negative HIV diagnostic test.
* Seronegative for hepatitis B surface antigen (HBsAg)
* Negative β-HCG (human chorionic gonadotropin) pregnancy test (urine or serum) on day of enrollment if woman is presumed to be of reproductive potential.
* For females only, willingness to practice continuous effective contraception (see section 6.4.3) during the study and a negative urine pregnancy test on the day(s) of screening and vaccination.

Exclusion Criteria:

* Recent exposure to Ebola virus infection (this is not a post-exposure vaccine)
* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Prior receipt of an investigational Ebola or Marburg vaccine, a chimpanzee adenovirus vectored vaccine, MVA vectored vaccine (for booster study) or any other investigational vaccine likely to impact on interpretation of the trial data
* Receipt of any live, attenuated vaccine within 28 days prior to enrolment
* Receipt of any subunit or killed vaccine within 14 days prior to enrolment
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, including urticaria, respiratory difficulty or abdominal pain
* Any history of hereditary angioedema, acquired angioedema, or idiopathic angioedema.
* Any history of anaphylaxis in reaction to vaccination
* Pregnancy, lactation or willingness/intention to become pregnant during the study
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition
* Poorly controlled asthma or thyroid disease
* Seizure in the past 3 years or treatment for seizure disorder in the past 3 years
* Bleeding disorder (eg. Factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venipuncture
* Any known history of cardiac disease (for the booster portion of the study only)
* Any other serious chronic illness requiring hospital specialist supervision
* Current anti-tuberculosis prophylaxis or therapy
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Suspected or known injecting drug abuse in the 5 years preceding enrolment
* Any clinically significant abnormal finding on screening biochemistry or hematology blood tests
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-09-27 (Actual); Study Completion 2016-09-27 (Actual)

PRIMARY OUTCOMES:
Solicited local reactogenicity - Number of participants with the specific outcome | For 7 days following each vaccination
  Occurrence of solicited local signs and symptoms following vaccination
Solicited systemic reactogenicity - Number of participants with the specific outcome | For 7 days following each vaccination
  Occurrence of solicited systemic signs and symptoms following vaccination

SECONDARY OUTCOMES:
Ebolavirus specific immunogenicity | At 7, 14, 28, 56, 112 and 168 days after vaccination. For those who participate in booster substudy, additional samples will be collected at these time points and no further samples would be timed from the priming dose
  ELISA and neutralization antigen-specific assays for antibody responses and intracellular cytokine staining assay for T cell responses after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Myrons M Levine, MD DTPH, Study Director — University of Maryland, Baltimore
Locations (1):
- Centre pour le Developpement des Vaccins - Mali, Bamako, Mali

IPD SHARING:
Plan to Share IPD: No